CLINICAL TRIAL: NCT00136877
Title: Effect of Tonsillectomy on Preventing Recurrent Streptococcal Throat Infections: A Randomized Controlled Trial
Brief Title: Tonsillectomy in Recurrent Tonsillitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oulu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diary nro 135/2001
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2006-12-29 (Estimated); Status verified 2006-12

CONDITIONS: Tonsillitis
Keywords: recurrent tonsillitis; streptococcus; tonsillectomy; prevention
MeSH Terms: conditions — Tonsillitis

INTERVENTIONS:
Procedure: (adeno)tonsillectomy

SUMMARY:
The purpose of this study is to determine whether tonsillectomy is effective in preventing further streptococcal pharyngitis episodes in patients with recurrent tonsillitis.

DETAILED DESCRIPTION:
Tonsillectomy is widely used worldwide in recurrent streptococcal tonsillitis, but its effect remains unknown.

In this randomized controlled trial, the effect of tonsillectomy (compared to watchful waiting) in preventing further culture proven symptomatic streptococcal pharyngitis episodes is studied. In addition, symptoms after the operation, side effects, and life quality issues are recorded.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 tonsillitis episodes during the preceding year (at least one verified by culture or antigen testing)

Exclusion Criteria:

* Other serious illness
* Long term antibiotic treatment for other disease
* Documented immunologic disorder
* Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2001-10; Study Completion 2005-12

PRIMARY OUTCOMES:
microbiologically confirmed streptococcal pharyngitis episodes

SECONDARY OUTCOMES:
side effects
symptoms
quality of life issues

CONTACTS AND LOCATIONS:
Overall Officials: Olli-Pekka Alho, MD, Study Director — Dept of Otolaryngology, University of Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Alho OP, Koivunen P, Penna T, Teppo H, Koskela M, Luotonen J. Tonsillectomy versus watchful waiting in recurrent streptococcal pharyngitis in adults: randomised controlled trial. BMJ. 2007 May 5;334(7600):939. doi: 10.1136/bmj.39140.632604.55. Epub 2007 Mar 8. PMID 17347187